CLINICAL TRIAL: NCT05654376
Title: Art Therapy to Promote Wellbeing and Self-care in Resident Physicians.
Acronym: ATMIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-ART-2022-21
Record Dates: First submitted 2022-11-23; First posted 2022-12-16 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Work-Related Stress
Keywords: Resident physician; Art therapy; Self-awareness; Sel-Care
MeSH Terms: conditions — Occupational Stress | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group art therapy (Experimental): Cycle of 6 2-hours bimonthly group art therapy sessions.
  Interventions: Behavioral: Art therapy

INTERVENTIONS:
Behavioral: Art therapy — Participant's creativity is stimulated by visual arts materials and various art therapy techniques, in relation to 6 topics: self-care, stress management, flourishing caregiving, challenging caregiving, loss and grief, and sense of professional meaning.
  The strategy consists of stimulating an observant and symbolic gaze, facilitating visual expression, promoting communication about what it has been expressed, and gather learning from the multidimensional impact of the creative art process (sensations, emotions, cognitions and spiritual experiences).

SUMMARY:
This study evaluates if an art therapy intervention could lower resident physician's work-related stress and if it could promote their self-care.

DETAILED DESCRIPTION:
The objective of this study is to determine if an art therapy intervention could promote the well-being of resident physicians of an university tertiary hospital, as specialized physicians trainees exposed to the risk of burnout.

Using a cycle of 6 bimonthly sessions of group art therapy, the intervention stimulates the creative activity of the participants through various art materials and techniques. Next, they are invited to share their reflexions about the artworks produced, with the group and in presence of the art therapist.

The study mainly evaluates the work-related stress and the self-care grade of the participants, before the intervention, just after it and after a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* belonging to the resident physicians collective of the Santa Creu i Sant Pau Hospital.

Exclusion Criteria:

* being with a diagnostic of major depression
* receiving psychotherapy o similar

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of a change in burnout level | From baseline assessed 1 week before art therapy sessions cycle starting, at 1 week after cycle completion.
  Score calculations from the validated Spanish version of the Maslach Burnout Inventory Test (MBI-GS). Minimum-maximum values of Exhaustion subscale: 0-54, lower scores mean better outcome; Minimum-maximum values of Cynicism subscale: 0-30, lower scores mean better outcome; Minimum-maximum values of Professional efficacy subscale: 0-48, lower scores mean worse outcome.
Assessment of a change in burnout level | From baseline assessed 1 week before art therapy sessions cycle starting, at 3 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Maslach Burnout Inventory Test (MBI-GS). Minimum-maximum values of Exhaustion subscale: 0-54, lower scores mean better outcome; Minimum-maximum values of Cynicism subscale: 0-30, lower scores mean better outcome; Minimum-maximum values of Professional efficacy subscale: 0-48, lower scores mean worse outcome.
Assessment of a change in burnout level | From baseline assessed 1 week before art therapy sessions cycle starting, at 6 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Maslach Burnout Inventory Test (MBI-GS). Minimum-maximum values of Exhaustion subscale: 0-54, lower scores mean better outcome; Minimum-maximum values of Cynicism subscale: 0-30, lower scores mean better outcome; Minimum-maximum values of Professional efficacy subscale: 0-48, lower scores mean worse outcome.

SECONDARY OUTCOMES:
Assessment of a change in work-related stress | From baseline assessed 1 week before art therapy sessions cycle starting, at 1 week after cycle completion.
  Score calculations from the validated Spanish version of the Perceived Stress Scale (PFS 14). Minimum-maximum values: 0-56; lower scores mean better outcome.
Assessment of a change in work-related stress | From baseline assessed 1 week before art therapy sessions cycle starting, at 3 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Perceived Stress Scale (PFS 14). Minimum-maximum values: 0-56; lower scores mean better outcome.
Assessment of a change in work-related stress | From baseline assessed 1 week before art therapy sessions cycle starting, at 6 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Perceived Stress Scale (PFS 14). Minimum-maximum values: 0-56; lower scores mean better outcome.
Assessment of a change in self-awareness | From baseline assessed 1 week before art therapy sessions cycle starting, at 1 week after cycle completion.
  Score calculations from the validated Spanish version of the Five Facet Mindfulness Questionnaire (FFMQ). Minimum-maximum values: 15-75; higher scores mean better outcome.
Assessment of a change in self-awareness | From baseline assessed 1 week before art therapy sessions cycle starting, at 3 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Five Facet Mindfulness Questionnaire (FFMQ). Minimum-maximum values: 15-75; higher scores mean better outcome.
Assessment of a change in self-awareness | From baseline assessed 1 week before art therapy sessions cycle starting, at 6 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Five Facet Mindfulness Questionnaire (FFMQ). Minimum-maximum values: 15-75; higher scores mean better outcome.
Assessment of a change in empathy | From baseline assessed 1 week before art therapy sessions cycle starting, at 1 week after cycle completion.
  Score calculations from the validated Spanish version of the Interpersonal Reactivity Index (IRI). Minimum-maximum values: 28-140, higher scores mean better outcome.
Assessment of a change in empathy | From baseline assessed 1 week before art therapy sessions cycle starting, at 3 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Interpersonal Reactivity Index (IRI). Minimum-maximum values: 28-140, higher scores mean better outcome.
Assessment of a change in empathy | From baseline assessed 1 week before art therapy sessions cycle starting, at 6 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Interpersonal Reactivity Index (IRI). Minimum-maximum values: 28-140, higher scores mean better outcome.
Assessment of a change in compassion | From baseline assessed 1 week before art therapy sessions cycle starting, at 1 week after cycle completion.
  Score calculations from the validated Spanish version of the Compassion and Satisfaction Fatigue Test (ProQoL version IV). Minimum-maximum values in each subscale: 10-50; Compassion satisfaction subscale: higher scores mean better outcome; Burnout subscale: higher scores mean a worse outcome; Secondary traumatic stress subscale: higher scores mean a worse outcome.
Assessment of a change in compassion | From baseline assessed 1 week before art therapy sessions cycle starting, at 3 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Compassion and Satisfaction Fatigue Test (ProQoL version IV). Minimum-maximum values in each subscale: 10-50; Compassion satisfaction subscale: higher scores mean better outcome; Burnout subscale: higher scores mean a worse outcome; Secondary traumatic stress subscale: higher scores mean a worse outcome.
Assessment of a change in compassion | From baseline assessed 1 week before art therapy sessions cycle starting, at 6 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Compassion and Satisfaction Fatigue Test (ProQoL version IV). Minimum-maximum values in each subscale: 10-50; Compassion satisfaction subscale: higher scores mean better outcome; Burnout subscale: higher scores mean a worse outcome; Secondary traumatic stress subscale: higher scores mean a worse outcome.
Assessment of a change in professional quality of life | From baseline assessed 1 week before art therapy sessions cycle starting, at 1 week after cycle completion.
  Score calculations from the validated Spanish version of the Professional Quality of Life Scale. Minimum-maximum values: 9-45; lower scores mean better outcome.
Assessment of a change in professional quality of life | From baseline assessed 1 week before art therapy sessions cycle starting, at 3 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Professional Quality of Life Scale. Minimum-maximum values: 9-45; lower scores mean better outcome.
Assessment of a change in professional quality of life | From baseline assessed 1 week before art therapy sessions cycle starting, at 6 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Professional Quality of Life Scale. Minimum-maximum values: 9-45; lower scores mean better outcome.
Assessment of a change in self-care | From baseline assessed 1 week before art therapy sessions cycle starting, at 1 week after cycle completion.
  Score calculations from the validated original Spanish version of Self-care Scale. Minimum-maximum values: 9-45; higher scores mean better outcome.
Assessment of a change in self-care | From baseline assessed 1 week before art therapy sessions cycle starting, at 3 months follow up after cycle completion.
  Score calculations from the validated original Spanish version of Self-care Scale. Minimum-maximum values: 9-45; higher scores mean better outcome.
Assessment of a change in self-care | From baseline assessed 1 week before art therapy sessions cycle starting, at 6 months follow up after cycle completion.
  Score calculations from the validated original Spanish version of Self-care Scale. Minimum-maximum values: 9-45; higher scores mean better outcome.
Assessment of a change in fear of death | From baseline assessed 1 week before art therapy sessions cycle starting, at 1 week after cycle completion.
  Score calculations from the validated Spanish version of the Collett-Lester Fear of Death Scale. Minimum-maximum values in each subscale: 7-35; higher scores mean worse outcome.
Assessment of a change in fear of death | From baseline assessed 1 week before art therapy sessions cycle starting, at 3 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Collett-Lester Fear of Death Scale. Minimum-maximum values in each subscale: 7-35; higher scores mean worse outcome.
Assessment of a change in fear of death | From baseline assessed 1 week before art therapy sessions cycle starting, at 6 months follow up after cycle completion.
  Score calculations from the validated Spanish version of the Collett-Lester Fear of Death Scale. Minimum-maximum values in each subscale: 7-35; higher scores mean worse outcome.

OTHER OUTCOMES:
Qualitative aspects gathered from the intervention | At 1 week after art therapy sessions cycle completion.
  Information gathered through a semi-structured questionnaire produced by the research team, about perceived helpfulness, emotions and sensations, preferences and drawbacks, learnings, expectation of a professional and/or personal impact.
Qualitative aspects gathered from the intervention | At 3 months follow up after art therapy sessions cycle completion.
  Information gathered through a semi-structured questionnaire produced by the research team, about perceived helpfulness, emotions and sensations, preferences and drawbacks, learnings, expectation of a professional and/or personal impact.
Qualitative aspects gathered from the intervention | At 6 months follow up after art therapy sessions cycle completion.
  Information gathered through a semi-structured questionnaire produced by the research team, about perceived helpfulness, emotions and sensations, preferences and drawbacks, learnings, expectation of a professional and/or personal impact.
Perception of a change process | At 1 week after art therapy sessions cycle completion.
  Audio recording interview and verbatim transcription to explore a possible experience of a change process.
Perception of a change process | At 3 months follow up after art therapy sessions cycle completion.
  Audio recording interview and verbatim transcription to explore a possible experience of a change process.
Perception of a change process | At 6 months follow up after art therapy sessions cycle completion.
  Audio recording interview and verbatim transcription to explore a possible experience of a change process.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pascual López, MD, Principal Investigator — Santa Creu i Sant Pau Hospital, Palliative Care Unit Director.
Locations (1):
- Hospital Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No